CLINICAL TRIAL: NCT04352894
Title: Indocyanine Green Fluorescence Detection of Peritoneal Carcinomatosis During Staging Laparoscopy for Gastric Cancer: Protocol for a Prospective Multicentric Single Arm Study
Brief Title: Intraoperative ICG Fluorescence Imaging for Peritoneal Carcinomatosis Detection
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia (Other)
Responsible Party: Principal Investigator, Gian Luca Baiocchi, Associate Professor, Azienda Socio Sanitaria Territoriale degli Spedali Civili di Brescia
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: AOBrescia_baiocchi_ICG1
Record Dates: First submitted 2020-04-14; First posted 2020-04-20 (Actual); Last update posted 2020-04-20 (Actual); Status verified 2020-04

CONDITIONS: Peritoneal Carcinomatosis; Gastric Cancer
MeSH Terms: conditions — Peritoneal Neoplasms; Stomach Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- fluorescence guided peritoneal exploration (Experimental): Indocyanine green (ICG) intravenous injection and peritoneal exploration with technology able to detect fluorescence generated by ICG
  Interventions: Diagnostic Test: Fluorescence guided peritoneal exploration

INTERVENTIONS:
Diagnostic Test: Fluorescence guided peritoneal exploration — Intravenous injection of ICG

SUMMARY:
Background. Peritoneal carcinomatosis is a frequent and deadly localization of gastric cancer. Available imaging techniques have a low accuracy in detecting small peritoneal nodules, and direct laparoscopic visualization may fail too. A more accurate staging technique would be advantageous for individualization of therapeutic path. Indocyanine Green (ICG) fluorescence imaging has been reported as a tool for visualizing small peritoneal seedings due to the "enhanced permeability and retention" (EPR) effect of cancer nodules.

Aim. To explore the feasibility and effectiveness of fluorescence-enhanced peritoneal carcinomatosis detection in patients with gastric cancer undergoing staging laparoscopy.

Methods. This prospective, multicentric, single arm study will include patients with gastric cancer, without a radiological suspicion of peritoneal carcinomatosis, undergoing staging laparoscopy. An intravenous injection of ICG is given at different dosage and at different timepoints before the intervention. During the staging laparoscopy, the abdominal cavity exploration is performed using standard white-light, and subsequently using fluorescence imaging. Suspicious nodules are harvested, until a maximum of 5 per patient, and sent for definitive histological examination. Peritoneal washing is also harvested for cytologic assessment in all cases. The eventual benefit of fluorescence imaging in terms of additional peritoneal lesions that were not detected during standard white-light imaging is evaluated.

Discussion. This study will establish if fluorescence imaging increases sensitivity and/or specificity of staging laparoscopy in detecting peritoneal carcinomatosis from gastric cancer. Improved accuracy may translate in better care path selection.

ELIGIBILITY:
Inclusion Criteria:

1. Age of ≥18years
2. Ability to provide written informed consent
3. Histologically confirmed gastric adenocarcinoma or oesophago-gastric junction adenocarcinoma Siewert 2 and 3
4. cT>1
5. cM0 (clinical staging: no metastases)
6. Staging laparoscopy is indicated by the internal work-up protocol
7. Staging laparoscopy is in accordance with NCCN (National Comprehensive Cancer Network) guidelines

Exclusion Criteria:

1. Pregnancy
2. Iodine allergy/sensibility
3. Clinical P1 (defined as high probability of peritoneal carcinomatosis at imaging)
4. Investigator judgement that the patient should not participate for any reason

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2020-09 (Estimated); Primary Completion 2021-09 (Estimated); Study Completion 2021-09 (Estimated)

PRIMARY OUTCOMES:
Best modality of ICG injection | intra-operative assessment
  best timing of injection

SECONDARY OUTCOMES:
Sensitivity of ICG fluorescence | intra-operative assessment
  As compared with white light

CONTACTS AND LOCATIONS:
Overall Officials: Gian Luca Baiocchi, Prof, Principal Investigator — ASST Spedali Civili, University of Brescia

IPD SHARING:
Plan to Share IPD: No